CLINICAL TRIAL: NCT04262999
Title: Assessment of Bone Mineral Density and Periodontal Status in Patients With Epilepsy on Mono- and Combination Therapy of Antiepileptic Drug: A Cross-sectional Study.
Brief Title: Bone Mineral Density and Periodontal Status in Patients on Antiepileptic Drug
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Other Study IDs: Swati perio
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- drug sodium valproate: individuals on antiepileptic drug sodium valproate for at least 1 year at the time of participation of the study.
  Interventions: Other: effect of sodium valproate on alveolar bone level
- drug levetiracetam: individuals on antiepileptic drug levetiracetam monotherapy for at least 1 year at the time of participation of the study.
  Interventions: Other: effect of levetiracetam on alveolar bone level
- drug sodium valproate + levetiracetam: individuals on antiepileptic drug sodium valproate + levetiracetam combination therapy for at least 1 year at the time of participation of the study.
  Interventions: Other: effect of sodium valproate+levetiracetam on alveolar bone level
- control group: systemically healthy individuals
  Interventions: Other: control group

INTERVENTIONS:
Other: effect of sodium valproate on alveolar bone level — Comparative evaluation of bone mineral density and levels of marginal alveolar bone in patients with epilepsy on sodium valproate drug therapy.Comparative evaluation of periodontal parameters in all the patients who are on sodium valproate drug therapy.
  Groups: drug sodium valproate
Other: effect of levetiracetam on alveolar bone level — Comparative evaluation of bone mineral density and levels of marginal alveolar bone in patients with epilepsy on levetiracetam drug therapy.Comparative evaluation of periodontal parameters in all the patients who are on levetiracetam drug therapy.
  Groups: drug levetiracetam
Other: effect of sodium valproate+levetiracetam on alveolar bone level — Comparative evaluation of bone mineral density and levels of marginal alveolar bone in patients with epilepsy on sodium valproate+levetiracetam drug therapy.Comparative evaluation of periodontal parameters in all the patients who are on sodium valproate+ levetiracetam drug therapy.
  Groups: drug sodium valproate + levetiracetam
Other: control group — Control group individuals will be systemically healthy.
  Groups: control group

SUMMARY:
Assessment of bone mineral density and periodontal parameters in patients with epilepsy. Comparative evaluation of bone mineral density and levels of marginal alveolar bone in patients with epilepsy on monotherapy, combination therapy, and systemically healthy individuals.Comparative evaluation of periodontal parameters in all the patients who are on monotherapy and combination therapy and in systemically healthy individuals.

DETAILED DESCRIPTION:
Epilepsy is one of the most commonly encountered neurological conditions. Approximately one-third of the patients affected by this disease need to have life-long treatment with antiepileptic drugs(AEDs) . Various studies have shown that AEDs are major risk factors for bone diseases not only in institutionalized individuals and those having low Vitamin-D consumption, reduced sunlight exposure and diminished physical activity but also in non-institutionalized patients, well-nourished ambulatory adults, postmenopausal women, older men and children with this disease.The earliest reports regarding the negative effect of antiepileptic drugs on bone metabolism date back to the late 1960s. Various studies have been performed to explore the relationship between AEDs and bone metabolism but findings remain inconclusive.

AEDs are given as either monotherapy or polytherapy. In monotherapy, the antiepileptic drugs which are most commonly associated with altered bone metabolism include carbamazepine, phenytoin, primidone and phenobarbitone. New generation AEDs such as lamotrigine(LTG), topiramate, levetiracetam(LEV) are approved to be used as both antiepileptic monotherapy as well as adjuvants in combination with other AEDs. Some studies showed a negative influence of these new AEDs on bone health while other studies reported contradictory findings.

Biochemical indices are used for the measurement of blood concentration of calcium ,phosphorus, vitamin D, parathyroid hormone,bone remodelling markers like receptor activator of nuclear factor-kappa B ligand (RANKL) and osteoprotegerin(OPG). All these markers identify the patients with bone disease in an indirect way. Bone mineral density (BMD) tests have utility in detecting osteoporosis, assessing risk for bone fracture and also monitoring the response to osteoporosis therapy. Values of BMD test depend upon bone mineral content(BMC) and bone size. Dual-energy x-ray absorptiometry (DEXA) is a painless, non-invasive and easy to use technique for detection of bone mineral density (BMD) with the added benefit of low radiation exposure. It was earlier demonstrated that AEDs possess the property of enzyme induction activity through hepatic cytochrome P450 enzyme system, and this was held causative for metabolic bone diseases by increasing vitamin D metabolism, secondary type hypocalcemia and hyperparathyroidism. However, various studies have reported that both non-enzyme inducing and enzyme inducing AEDs have the potential to result in metabolic bone disease.

R.A. Seymour et al. (1985) conducted a study in which they investigated the periodontal health of adult patients with epilepsy matched in two groups and treated with either sodium valproate or phenytoin drug therapy. They reported that significantly less bone loss was observed in the phenytoin group than those on sodium valproate or the control patients. The limitation of this study was a small sample size and selection of anterior teeth only for recording periodontal parameters and alveolar bone loss.

The present study has been designed with the aim to compare bone mineral density, periodontal parameters and marginal alveolar bone levels in individuals who are on antiepileptic drugs - either sodium valproate or levetiracetam as monotherapy or on a combination regime of both the drugs(sodium valproate and levetiracetam) for at least 1 year with systemically healthy individuals. The present cross-sectional study will be conducted in the Department of periodontology, Post Graduate Institute of Dental Sciences, Rohtak in collaboration with Department of neurology, Post Graduate Institute of Medical Sciences, Rohtak.

STUDY PERIOD- January 2020 to April 2021 SAMPLE SIZE- A sample size of total 140 participants was calculated by using basic formula of sample size calculation with an moderate effect size 0.3,alpha =0.05 and power=0.80.The cross-sectional study will include 140 individuals, who will be comprised into 4 groups and the individuals in each group will be recruited as Test group 1 - individuals on antiepileptic drug sodium valproate for at least 1 year at the time of participation of the study.Test group 2- individuals on antiepileptic drug levetiracetam monotherapy for at least 1 year at the time of participation of the study.Test group 3 - individuals on antiepileptic drug sodium valproate + levetiracetam combination therapy for at least 1 year at the time of participation of the study.Control group- systemically healthy individuals.Dose of AEDs would be adjusted by treating neurologist as per the clinical response to achieve adequate seizure control.Patients in test group will be recruited from the Outpatient Department of Neurology, Post Graduate Institute of Medical Sciences, Rohtak.Patients in control group will be recruited from Department of Oral Medicine and Radiology, Post Graduate Institute of Dental Sciences, Rohtak.TEST GROUP AND CONTROL GROUP - Periodontal parameters:- 1.PLAQUE INDEX(PI) 2.GINGIVAL INDEX (GI) 3. BLEEDING ON PROBING (BOP) 4.PROBING POCKET DEPTH (PPD): 5. CLINICAL ATTACHMENT LEVEL (CAL) 6. BODY MASS INDEX (BMI) 7.CDC-AAP CASE DEFINIATIONS FOR SURVEILLANCE OF PERIODONTITIS46

1. No periodontitis- No evidence of mild, moderate, or severe periodontitis
2. Mild periodontitis- ≥2 interproximal sites with AL ≥3 mm, and ≥ 2 interproximal sites with PD ≥4 mm (not on same tooth) or one site with PD ≥5 mm
3. Moderate periodontitis- ≥2 interproximal sites with AL ≥4 mm (not on same tooth), or ≥2 interproximal sites with PD ≥5 mm (not on same tooth)
4. Severe periodontitis- ≥2 interproximal sites with AL ≥6 mm (not on same tooth) and ≥1 interproximal site with PD ≥5 mm (Third molars will be excluded; total periodontitis is deﬁned as the sum of mild, moderate, and severe disease Radiographic parameters:-1.DUAL ENERGY X-RAY ABSORPTIOMETRY (DEXA) 2.RADIO-VISIOGRAPHY (RVG)

ELIGIBILITY:
Inclusion Criteria:

* Individuals will be included in the study with the age range of 18-40 years. The selection of individuals will be according to age group, body mass index, and duration of drug therapy.

Control group individuals will be systemically healthy. Test group individuals will comprise of individuals diagnosed with epilepsy according to the International League Against Epilepsy (ILAE) criteria,1981 and monitored by the Department of Neurology, Post Graduate Institute of Medical Sciences, Rohtak.

The duration of antiepileptic drugs should at least 1 year at the time of enrollment.

Exclusion Criteria: Post-menopausal women The disease that affect bone health like Paget's disease, Multiple myelomas, osteoporosis.

Individuals who are already taking steroid therapy, Bisphosphonates therapy. Individuals on vitamins and calcium supplements. With a history of substance abuse (Tobacco/Alcohol) Malabsorption syndrome (Ulcerative colitis, Crohn's disease, Celiac disease, etc.)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients in the test group will be recruited from the Outpatient Department of Neurology, Post Graduate Institute of Medical Sciences, Rohtak.
  Patients in the control group will be recruited from the Department of Oral Medicine and Radiology, Post Graduate Institute of Dental Sciences, Rohtak.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | 1year
  DUAL ENERGY X-RAY ABSORPTIOMETRY (DEXA)- There are two s.d. scores, T-scores and Z-scores. The T-scores compare the BMD values obtained with a sex-matched and race matched population at peak BMD, while the Z-scores compare the BMD measurements with an age-matched population. According to the WHO, patients with scores that are 1 - 2.5 s.d. below normal DEXA-values have osteopenia, while those with values >2.5 s.d. below normal values are described as osteoporotic. When evaluating DEXA scans, 1 s.d. represents a T-score of 1. Thus, a patient with an s.d. of 3 below normal (i.e., osteoporosis) will have a T-score of -3.
Marginal alveolar bone levels | 1 year
  By using RVG with the help of XCP-film holder, levels of marginal bone will be measured from Cemento-enamel junction to crest of alveolar bone on mesial and distal aspect of index teeth (first molar of each quadrant and central and lateral incisors of 2nd and 4th quadrant) Index teeth for scoring will be 1st molar from each quadrant and central and lateral incisor of 2nd and 4th quadrant. If index teeth are missing then we will take adjacent teeth as index teeth in our study.

SECONDARY OUTCOMES:
Plaque Index (PI) | 1year
  Plaque index by Silness and Loe(1964) will be used for assessment of plaque. For the scoring, a mouth mirror, an explorer and a light source will be used on air dried teeth and gingiva. Criteria for recording the scores will be as follows.
  SCORE CRITERIA 0 No plaque
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque could only be recognised by running a probe across the tooth surface area
  2. Moderate accumulation of soft deposits within the gingival pocket, or the tooth and gingival margin, which can be seen with the naked eyes.
  24
  3 Abundance of soft matter on tooth and/or on the gingival margin.
Gingival Index (GI) | 1year
  Gingival Index by Loe and Silness (1963) will be used for assessment of severity of gingival inflammation. For the scoring, a mouth mirror, a probe and a light source will be used on air dried teeth and gingiva. Criteria for recording the scores:
  Score Criteria 0 Absence of inflammation/normal gingiva.
  1. Mild inflammation, slight change in colour, slight oedema; no bleeding on probing within 30 seconds.
  2. Moderate inflammation; moderate glazing, redness, oedema, hypertrophy and bleeding on probing.
  3. Severe inflammation; marked redness and hypertrophy ulceration of gingival margin. Tendency to spontaneous bleeding.
  Diagnosis of gingivitis will be assigned when BOP was present at >50% of all sites and PD was <3 mm at ≥90% of the measured sites but ≤1 site had PD >4 mm and CAL≤1 mm and no clinical and/or radiographic sign of periodontitis will be evident.
Bleeding On Probing (BOP) | 1year
  BOP will be recorded as 1 (present) if it occurred within 15 sec of probing and 0 (absent) if no bleeding occurred. It will be calculated in %. After adding all the scores, total score will be divided by the total no. of surfaces accessed and multiplied by 100. It will be designed as % sites with bleeding on probing.
Pocket Probing Depth (PPD) | 1year
  Probing pocket depth will be measured as the distance from the gingival margin to the base of the clinical pocket. The probing depth measurements will be assessed using a calibrated manual periodontal probe (PCP-UNC 15 Hu-Friedy, Chicago, IL, USA). The probe will be inserted with a firm, gentle pressure to the bottom of the pocket and maintained parallel to the vertical axis of the tooth. Measurements will be noted at 6 sites of involved tooth - mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual. Measurements will be rounded to the nearest whole millimetre.
Clinical Attachment Loss (CAL) | 1year
  Clinical Attachment Level will be measured as the distance between the base of the clinical pocket and the cemento-enamel junction(CEJ).Measurements will be made at 6 sites of involved tooth- mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual using UNC-15 probe. Measurements will be rounded to the nearest whole millimetre. Distance of base of the pocket from gingival margin, distance of free gingival margin from CEJ.

CONTACTS AND LOCATIONS:
Overall Officials: Swati Jaglan, MDS, Principal Investigator — Post Graduate Institute of Dental Sciences,Rohtak
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
Study protocol
Supporting Information: Study Protocol